CLINICAL TRIAL: NCT05499754
Title: The Effect of Supralottic Airway Devicess on Hemodynamic Response and Optic Nerve Sheath Diameter. PROSEAL LMA, SUPREMA LMA, I-JEL LMA
Brief Title: Effect of Different Supralottic Airway Devicess on Optic Nerve Sheath Diameter
Status: Completed | Type: Observational
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Gamze Küçükosman, medical doctor, Zonguldak Bulent Ecevit University
Other Study IDs: 2019/09
Record Dates: First submitted 2022-06-02; First posted 2022-08-12 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Intracranial Pressure Increase; Supraglottic Airway Device; Optic Nerve Sheath Diameter
Keywords: Supraglottic airway device; hemodynamic response; optic nerve sheath diameter
MeSH Terms: conditions — Intracranial Hypertension

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- pLMA(n=30)
  Interventions: Other: pLMA: PROSEAL LARYNGEAL MASK, sLMA : SUPREMA LARYNGEAL MASK, I-jel =I-GEL
- sLMA(n=30)
  Interventions: Other: pLMA: PROSEAL LARYNGEAL MASK, sLMA : SUPREMA LARYNGEAL MASK, I-jel =I-GEL
- I-jel(n=30)
  Interventions: Other: pLMA: PROSEAL LARYNGEAL MASK, sLMA : SUPREMA LARYNGEAL MASK, I-jel =I-GEL

INTERVENTIONS:
Other: pLMA: PROSEAL LARYNGEAL MASK, sLMA : SUPREMA LARYNGEAL MASK, I-jel =I-GEL — a SAD was inserted by all anaesthetists participating in the study had at least 3 years experience of airway management and were experienced with both the pLMA, sLMA and I-jel. Inadequate ventilation after two attempts was considered a failed placement, and these patients were excluded, while the practitioner was freed to use an alternative airway device.

SUMMARY:
Direct laryngoscopy and tracheal intubation are associated with increases in intraocular pressure (IOP), intracranial pressure (ICP), heart rate (HR), and blood pressure. The use of supraglottic airway devices (SADs) are known to be beneficial in overcoming the disadvantages of laryngoscopy and tracheal intubation, especially ocular and pressure stress responses. In recent years, it has been reported that ultrasonographic measurement of optic nerve sheath diameter (ONSD) can be used in the diagnosis of increased ICP. The aim of our study is to compare the effects of Proseal laryngeal mask airway (pLMA), Suprem laryngeal mask airway (sLMA) and I-gel on hemodynamic response and ONSD during insertion in adult patients.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status of I-II
* elective surgery
* non-ophthalmic procedures
* 1-2 h duration
* general anaesthesia
* supine position

Exclusion Criteria:

* Mallampati and ASA status ≥III,
* a history or suspect of difficult airway,
* previous intracranial/ocular surgery,
* cerebral edema/high intracranial pressure,
* glaucoma,
* uncontrolled hypertension

  -, diabetic retinopathy,
* obstetric patients,
* those who refused to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 90
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
OPTIC NERVE SHEATH DIAMETER | 10 min after using supraglottic airway devices
  effects of different types of laryngeal masks onoptic nerve sheath diameter

CONTACTS AND LOCATIONS:
Locations (1):
- Gamze Küçükosman, Zonguldak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No